CLINICAL TRIAL: NCT07083453
Title: Financial Incentives to Encourage Uptake of Preventive Dental Care Services Among Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Tan Hui Xuan Sharon, Research Fellow, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NUS-IRB-2023-49
Record Dates: First submitted 2025-07-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Dental
Keywords: Dental care; Oral health; Economics; Reimbursement; Incentive; Patient acceptance of health care
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Active Comparator): $10 rebate offered
  Interventions: Other: Control
- Comparator 1 (Active Comparator): $10 rebate offered with online and caries risk assessment
  Interventions: Other: Comparator 1
- Comparator 2 (Active Comparator): $20 rebate offered
  Interventions: Other: Comparator 2
- Comparator 3 (Active Comparator): $30 rebate offered
  Interventions: Other: Comparator 3
- Comparator 4 (Active Comparator): $50 rebate offered
  Interventions: Other: Comparator 4

INTERVENTIONS:
Other: Comparator 1 — $10 rebate offered with an online caries and periodontal risk assessment
  Arms: Comparator 1
Other: Comparator 2 — 20 rebate offered without risk assessment
  Arms: Comparator 2
Other: Comparator 3 — $30 rebate offered without risk assessment
  Arms: Comparator 3
Other: Comparator 4 — $50 rebate offered without risk assessment
  Arms: Comparator 4
Other: Control — $10 rebate offered with no risk assessment
  Arms: Control

SUMMARY:
The study aims to assess if financial rebates affect the uptake of dental services among adults, determine the optimal level of financial rebates to encourage dental visits, and assess the factors associated with the uptake of dental services.

DETAILED DESCRIPTION:
Aim:

The project aims to assess the effect of various factors on the uptake of preventive dental services, including the impact of out-of-pocket costs on the uptake of preventive dental services.

The hypotheses of the study are:

1. Out-of-pocket costs affect the uptake of preventive dental services
2. A financial subsidy covering at least 50% of costs would increase the uptake of preventive dental services
3. Financial subsidies have a greater impact on dental utilization among low-income adults compared to high income adults

ELIGIBILITY:
Inclusion Criteria:

* Between 21 and 85 years of age (inclusive)
* Able to provide informed consent to participate in the study
* Able to read and comprehend English

Exclusion Criteria:

* Individuals with cognitive impairments or mental health conditions

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5500 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of dental services | From baseline to up to 2 years after intervention
  Uptake of dental services

SECONDARY OUTCOMES:
Change in oral hygiene practices | From baseline to 1 year after intervention
  Change in % of participants that brush their teeth at least twice a day
Change in dietary practices | From baseline to 1 year after intervention
  Change in % of participants that consume sugary foods or drinks at least once a day
Change in oral health related quality of life | From baseline to 1 year after intervention
  Change in Oral Health Impact Profile-14 (OHIP-14) score. Minimum score: 0, Maximum score: 56. Higher scores reflect a worse outcome
Change in quality of life | From baseline to 1 year after intervention
  Change in EuroQol five-dimension, five-level (EQ-5D-5L) score. Health states range from 11111 (best possible health state) to 55555 (worst possible health state).

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed pending participant consent.